CLINICAL TRIAL: NCT01476020
Title: Is There A LIfe for DES After Discontinuation of Clopidogrel:The ITALIC PLUS Trial
Brief Title: Is There A LIfe for Drug Eluting Stent (DES) After Discontinuation of Clopidogrel
Acronym: ITALICplus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gilard, Martine (Individual)
Collaborators: Clinical Research Organization and study management (Unknown); Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011 08
Record Dates: First submitted 2011-11-03; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Restenosis
Keywords: Drug eluting stent; Dual antiplatelet therapy; bleeding; stent thrombosis; follow-up of the drug eluting stent
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- no clopidogrel 6 months after DES: Patients with a single treatment antiplatelet therapy (aspirin) 6 months after drug-eluting stent implantation (Xience V Abbott company), including a 12-, 24- and 36-month follow-up analysis.
- 2 antiplatelet therapy 2 years after DES: patients with dual antiplatelet therapy with clopidogrel and aspirin 24 months after drug-eluting stent implantation, including a 12-, 24- and 36-month follow-up analysis.

SUMMARY:
The ITALIC PLUS Trial was designed with the objective of extending to other countries the enrollment of patients into the ITALIC trial initially conducted in France, in order to achieve statistical significance by pooling the data of both trials.

DETAILED DESCRIPTION:
The use of drug-eluting stents has resulted in a significant reduction in the restenosis rate and in the need for repeat angioplasty of the stented lesion. However, the occurrence of late stent thrombosis has resulted in an increase in the duration of dual antiplatelet treatment.

According to the guidelines of the ESC, the current recommended duration of dual antiplatelet treatment is 12 months.

A relationship has been demonstrated between the occurrence of late stent thrombosis and aspirin resistance.

Furthermore, dual anti-platelet treatment is associated with an increase in bleeding, the severity of which has been well documented. In addition, the patients involved, and especially those over 70, have significant co-morbidities often requiring extra-cardiac surgery which cannot easily be carried out in patients on dual antiplatelet treatment or clopidogrel.

The objective of this study is to determine whether, after a period of 6 months following Drug eluting stent (DES) implantation in patients regarded as sensitive to aspirin, dual antiplatelet therapy may be replaced by aspirin alone.

The original Italic Trial is a multicenter, randomized study evaluating the non-inferiority of aspirin as a single treatment versus dual antiplatelet therapy with clopidogrel and aspirin 6 months after drug-eluting stent implantation, including a 12-, 24- and 36-month follow-up analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥ 18 years of age eligible for PCI with at least one drug eluting stent (name: Xience) implanted in all clinical situations excluding primary PCI for acute MI and treatment of the left main artery.
* Male or female subject ≥ 18 years of age eligible for PCI with at least one DES Xience.
* Patient not pre-treated with protein IIb/IIIa inhibitors (name: abxicimab or eptifibatide) during hospitalization
* Patient pre-treated with aspirin and clopidogrel before PCI
* ASA check at least 24 hours after the interruption of tirofiban
* The subject has given written informed and dated consent to participate in this study.

Exclusion Criteria:

* Subjects not able to give informed consent
* Prior implantation of DES
* Known platelets < 100 000/µl or known hemorrhagic diathesis
* Oral anticoagulation or treatment with abxicimab or eptifibatide during hospitalization
* ASA check less than 24 hours after the interruption of tirofiban
* Thrombolytic therapy within 4 days before ASA check
* Contra-indication to aspirin or clopidogrel
* Recent major surgery < 6 weeks
* Evidence of an active gastrointestinal or urogenital bleeding
* Severe liver insufficiency
* Primary PCI for acute MI
* Left main PCI
* Any scheduled surgery during the year after enrollment
* Severe concomitant disease with life expectation < two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are selected from the general population needing Percutaneous Coronary Interventions (PCI).
Sampling Method: Probability Sample
Enrollment: 1240 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
composite endpoint:death, myocardial infarction, repeat angioplasty due to the occurrence of restenosis, occurrence of stroke and major bleeding | one year

SECONDARY OUTCOMES:
composite endpoint:Death, myocardial infarction, repeat angioplasty due to the occurrence of restenosis, occurrence of stroke and major bleeding and minor bleeding | 36-month period

CONTACTS AND LOCATIONS:
Overall Officials: martine Gilard, MD,PhD, Principal Investigator — Brest University France
Locations (1):
- Department of cardiology, Brest, France

REFERENCES:
- [Derived] Gilard M, Barragan P, Noryani AAL, Noor HA, Majwal T, Hovasse T, Castellant P, Schneeberger M, Maillard L, Bressolette E, Wojcik J, Delarche N, Blanchard D, Jouve B, Ormezzano O, Paganelli F, Levy G, Sainsous J, Carrie D, Furber A, Berland J, Darremont O, Le Breton H, Lyuycx-Bore A, Gommeaux A, Cassat C, Kermarrec A, Cazaux P, Druelles P, Dauphin R, Armengaud J, Dupouy P, Champagnac D, Ohlmann P, Endresen K, Benamer H, Kiss RG, Ungi I, Boschat J, Morice MC. 6- versus 24-month dual antiplatelet therapy after implantation of drug-eluting stents in patients nonresistant to aspirin: the randomized, multicenter ITALIC trial. J Am Coll Cardiol. 2015 Mar 3;65(8):777-786. doi: 10.1016/j.jacc.2014.11.008. Epub 2014 Nov 16. PMID 25461690